CLINICAL TRIAL: NCT06677515
Title: Improving Social Functioning in People With Substance Use and Mental Health Disorders Using Virtual Reality (ROPVR): Study Protocol for a Multi-centre, Pragmatic Randomized Controlled Trial
Brief Title: Improving Social Functioning in People With Substance Use and Mental Health Disorders Using VR
Acronym: ROPVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 326773VR_WP3
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Mental Disorder
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) training (Experimental): Participants randomized to the intervention arm will attend VR sessions twice a week in 5 weeks, or 10 sessions in total. They will be placed into different virtual environments with increasing complexity, where they will be confronted with normal everyday situations in city environments.
  In the first session, participants will receive instructions on using the head mounted display and navigating the scenarios. In three scenarios, participants are only observers, while in the remaining they can choose between several response options. These responses will be displayed on the screen, and participants can select their preferred response by pointing their finger to the chosen response alternative. The response alternatives are also provided verbally.
  Interventions: Other: VR training
- Treatment as usual (No Intervention): Treatment of substance use disorders (SUD) is delivered by personnel with medical, psychological, and social expertise, meeting specialist-level healthcare standards. SUD treatment clinics offer patient-centred, interdisciplinary, holistic treatment focusing on physical, mental and social problems. Treatment often consists of both individual and group therapies and include activities (e.g., physical exercise, social activities) in the clinic as well as in external settings. Since treatment approaches and facilities may vary across clinics, patients' preferences or choice of clinic are emphasized. According to national guidelines, persons with SUD and co-occurring severe mental illness (i.e., schizophrenia or severe bipolar disorder) can receive treatment in SUD treatment clinics as long as their mental condition is stable. Otherwise, persons with SUD and severe mental illness receive treatment for both conditions within mental health services.

INTERVENTIONS:
Other: VR training — The different VR scenarios comprise the following learning goals: 1) Social cognition. Interpreting social situations, understanding others; 2) Social communication. Express oneself, being understood by others; 3) Social competence. Interacting with others The investigators will use an MSI Raider GE78HX with a GeForce RTX4080 12GB GPU, running Windows 11, Unreal Engine 5.4, and the Meta Quest Link app, with a Meta Quest Pro as a PCVR headset connected via a Meta Quest Link cable. The setup works 100% locally, and no Wi-Fi or internet connection is used on the head-mounted-display or PC. The VR program itself does not store any data and will discard all that has happened inside the program, when restarted.
  Other Names: Training, using a virtual reality goggles
  Arms: Virtual reality (VR) training

SUMMARY:
ROPVR, a multi-centre, pragmatic randomized controlled trial (RCT) aims to evaluate a VR-technology which has been developed within an exploratory study and a development study, which facilitates social functioning among persons with a substance use and mental health disorder. Investigators will test a VR-program versus treatment as usual among patients enrolled into a long-term addiction-treatment facility. The RCT aims to evaluate the effectiveness of VR training compared to treatment as usual in improving resilience, quality of life, practical and social functioning and social participation (from baseline to 6 months), and to evaluate the cost-effectiveness of VR training versus treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or older receiving in-patient SUD treatment in specialized addiction treatment units in South-East Norway. This may include persons serving prison sentences during in-patient treatment according to the Execution of Sentences Act in Norway
* having the capability to read, understand and sign the Norwegian informed consent form
* willing and able to attend VR training two times a week for 5 weeks

Exclusion Criteria:

* significant visual, auditory, or balance impairment or other diseases affecting safety during VR sessions (e.g., epilepsy)
* current clinically significant severe mental health disorder (e.g., acute episode of psychosis or current active suicidal plans). Persons with psychotic disorders or other severe mental illness are not excluded if their condition is stable.
* severe travel sickness as a proxy for simulation sickness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Health and disability | From enrolement into the study until ca. 6 month
  The primary outcome measure is disability measured with the 36-item WHO Disability Assessment Schedule (WHODAS 2.0) total score at 6 months post-intervention. WHODAS 2.0 measures health and disability in adults and captures the level of functioning in 6 domains: cognition, mobility, self-care, getting along, life activities and participation. The scores assigned to each of the items - "none" (1), "mild" (2) "moderate" (3), "severe" (4) and "extreme" (5) - are summed. Scores from each of the items are simply added up without recoding or collapsing of response categories; thus, there is no weighting of individual items. Higher sum score indicates more problems. WHODAS is based on the conceptual framework of the International Classification of Functioning. WHODAS is trans diagnostic, culturally sensitive and covers all diseases, including physical, mental and substance use disorders. It is is suitable for measuring the clinical effectiveness of interventions.

SECONDARY OUTCOMES:
Practical and social functioning | From enrolement into the study until ca. 6 month
  Measured by the Practical and Social Functioning Scale (PSF 3) consists of 32 items and 8 domains: personal hygiene, communication, managing economy, housekeeping, contact with social network, personal health care, transportation, and work and activities. Each item is rated on a five-point response scale from 1 (does not apply) to 5 (applies completely). Based on the completed form, scores for the different parts can be calculated as follows:
  Total score for the entire scale with 28 items (sum 28 - 140, average score 1.0 - 5.0) Subscales (sum for each subscale 5 - 20, average score 1.0 - 5.0) Dimension activity (16 items, sum 16 - 80, average score 1.0 - 5.0) Dimension participation (12 items, sum 12 - 60, average score 1.0 - 5.0
Social participation | From enrolement into the study until ca. 6 month
  Mini-SCOPE comprises 25 items and measures 5 domains of Satisfaction with Opportunities (SatOpps) in terms of leisure time, community involvement, work, finances and family; 2 domains of Perceived Opportunities (PerOpps) regarding housing and income. It also contains a question on the perceived level of overall social inclusion and a question on the perceived level of quality of life. Mini-SCOPE includes 17 scorable items, while 8 other items are either Yes/No questions or about basic demographics. The SatOpps items were measures on a 7-point scale, ranging from 'delighted' to 'terrible', while the PerOpps items were measures on a 5-point scale. SatOpps and PerOpps are scored by calculating the sum of the items. Overall social inclusion and quality of life are single items and are scored separately. In all scorable items, higher scores indicate lower satisfaction opportunities, perceived opportunities or satisfaction with social inclusion and quality of life.
Resilience | From enrolement into the study until ca. 6 month
  To measure resilience, the Connor-Davidson Resilience Scale, 10 item version (CD-RISC 10) will be used. The CD-RISC-10 consists of 10 statements describing different aspects of resilience. The scale serves mainly as a measure of hardiness, with items corresponding to flexibility (1 and 5), sense of self-efficacy (2, 4 and 9), ability to regulate emotion (10), optimism (3, 6 and 8) and cognitive focus/maintaining attention under stress (7). Each item is scored on a five-point scale ranging from 0 to 4, with 0 representing that the resilience statement is not at all true and a score of 4 indicating that the statement is true nearly all the time. The total score is obtained by adding up all 10 items. The total can therefore range from 0 to 40. Higher scores suggest greater resilience and lower scores suggest less resilience, or more difficulty in bouncing back from adversity.
Cost-effectiveness | From enrolement into the study until ca. 12 month
  Health state descriptions of the study participants will be measured by EQ-5D-5L at baseline (T0), T1, T2 and T3. The EQ-5D-5L is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. It comprises comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression). Healthcare resource use, will be assessed using The Treatment Inventory of Costs in Patients with Psychiatric Disorders (TIC-P).

CONTACTS AND LOCATIONS:
Overall Officials: Marja Leonhardt, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (2):
- Norway (2):
  - Innlandet Hospital Trust, Brumunddal
  - Sykehuset Innlandet HF, Hamar

IPD SHARING:
Plan to Share IPD: Undecided
As we are collecting sensitive data, we are by rules and regulations not allowed to share any data. However, we might consider sharing pseudonymized data gradually.

REFERENCES:
- See also: Project website - in Norwegian only — https://www.sykehuset-innlandet.no/fag-og-forskning/forskning/ropforsk/forskningsprosjekter/rop-vr/